CLINICAL TRIAL: NCT06177301
Title: A Phase III Clinical Study of Tislelizumab Combined With GX Regimen Versus Tislelizumab Combined With GP Regimen in the First-line Treatment of Recurrence or Metastasis (R/M) Nasopharyngeal Carcinoma (NPC)
Brief Title: Tislelizumab Plus GX Versus Tislelizumab Plus GP in the Treatment of R/M NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associated Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-NC-001
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with GX (Experimental): Patients will receive tislelizumab combined with GX regimen： Tislelizumab：200mg vgtt，q3w；treatment until disease progression, patients withdrawal of informed, or intolerable toxicity.
  Gemcitabine：1000mg/m2, vgtt, d1,8, q3w, repeat 4-6 cycles. Capecitabine: 1000mg/m2, bid，po, d1-14, q3; treatment until disease progression, patients withdrawal of informed, or intolerable toxicity.
  Interventions: Drug: Tislelizumab combined with GX
- Tislelizumab combined with GP (Experimental): Patients will receive tislelizumab combined with GX regimen： Tislelizumab: 200mg vgtt，q3w；treatment until disease progression, patients withdrawal of informed, or intolerable toxicity.
  Gemcitabine: 1000mg/m2, vgtt, d1,8, q3w, repeat 4-6 cycles； Cisplatin: 80mg/m2, ivgtt, d1 (high-dose cisplatin antiemetic and hydration regimen), q3w，repeat 4 ~ 6 cycles.
  Interventions: Drug: Tislelizumab combined with GP

INTERVENTIONS:
Drug: Tislelizumab combined with GX — Tislelizumab：200mg vgtt，q3w；treatment until disease progression, patients withdrawal of informed, or intolerable toxicity.
  Gemcitabine：1000mg/m2, vgtt, d1,8, q3w, repeat 4-6 cycles. Capecitabine: 1000mg/m2, bid，po, d1-14, q3; treatment until disease progression, patients withdrawal of informed, or intolerable toxicity.
  Arms: Tislelizumab combined with GX
Drug: Tislelizumab combined with GP — Tislelizumab: 200mg vgtt，q3w；treatment until disease progression, patients withdrawal of informed, or intolerable toxicity.
  Gemcitabine: 1000mg/m2, vgtt, d1,8, q3w, repeat 4-6 cycles； Cisplatin: 80mg/m2, ivgtt, d1 (high-dose cisplatin antiemetic and hydration regimen), q3w，repeat 4 ~ 6 cycles.
  Arms: Tislelizumab combined with GP

SUMMARY:
The study is being conducted to evaluate the safety and efficacy of tislelizumab combined with GX regimen versus tislelizumab combined with GP regimen in the first-line treatment of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological examination confirmed recurrence or metastasis of nasopharyngeal carcinoma;
2. Patients who have not previously received systemic treatment for recurrent or metastatic diseases (For patients who have previously received induction chemotherapy, adjuvant chemotherapy or concurrent chemoradiotherapy, patients who relapsed at least 6 months after the cessation of chemotherapy can be enrolled).
3. Age: 18-75 years old, male or female;
4. Perfomance Status: 0~1;
5. At least one measurable lesion (according to RECIST v1.1, long diameter of measurable lesion scanned by spiral CT should be ≥ 10 mm or short diameter of swollen lymph node should be ≥ 15 mm; according to RECIST vl.1 standards, a previously treated lesion with local treatment can be used as target lesions after clear progress);
6. Blood routine examination: 1) Hemoglobin (HB)≥ 90g / L; 2) Neutrophil count (ANC) ≥ 1.5 × 109 / L; 3) platelets (PLT) ≥ 80 × 109 / L;
7. Liver function: 1) Serum total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN); 2) alanine aminotransferase (ALT), aspartate aminotransferase (AST])< 2.5 × ULN; if liver metastasis, ALT and AST ≤ 5 × ULN; Renal function: Albumin ≥ 28g / L ；Serum creatinine (Cr) ≤ 1.5 × ULN，or creatinine clearance rate ≥ 60 ml / min ;
8. Coagulation function : APTT and international normalized ratio (INR)< 1.5 × UNL;
9. Patients of childbearing age agree to take appropriate contraceptive measures. Serum pregnancy test was negative in women of childbearing age within 2 weeks before enrollment.
10. Patients agree to provide pathological tissue specimens (wax blocks or paraffin tissue sections 5-10 pieces) ;
11. Expected survival ≥ 3 months;
12. Patients volunteered to participate in this study and signed informed consent;

Exclusion Criteria:

1. Patients with local recurrence and suitable for surgery or radiotherapy;
2. Patients with a known history of severe allergies to monoclonal antibody therapy;
3. Patients who had previously received PD-1 monoclonal antibody or PD-L1 monoclonal antibody or CTLA4 monoclonal antibody;
4. Clinical significance of heart disease, including severe cardiac insufficiency : New York Heart Association (NYHA) cardiac insufficiency grade IV, unstable angina, acute myocardial infarction within 6 months before screening, congestive heart failure, Q-Tc interval greater than 500ms;
5. Patients with autoimmune diseases requiring treatment, or patients with a history of systemic use of steroids / immunosuppressive agents, such as : hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism;
6. Other serious and uncontrollable concomitant diseases that may affect the compliance of the program or interfere with the interpretation of the results, including uncontrolled diabetes, or lung diseases (interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchial spasm) ;
7. Known hepatitis B (HBV) (HBsAg positive and HBV-DNA ≥ 103IU / ml), hepatitis C ( HCV) infection (HCV antibody positive and HCV-RNA measurable) ; and other subjects with acquired and congenital immunodeficiency diseases, including, but not limited to, those infected with HIV;
8. Severe active infection;
9. Symptomatic patients with central nervous system metastasis;
10. Patients with a history of other malignant tumors (unless those who have been cured for more than 5 years);
11. Have a serious history of neurological or psychiatric disorders, including dementia or epilepsy;
12. Drug abuse, medical, psychological or social conditions that may interfere with the participant 's participation in the study or the evaluation of the study results;
13. Researchers believe that patients who are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To compare the progression-free survival of tislelizumab combined with GX regimen and tislelizumab combined with GP regimen based on the ITT analysis set evaluated by the researchers according to RECIST v1.1. | up to approximately 3 years
  Time from the date of enrollment to of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.

SECONDARY OUTCOMES:
To compare the objective response rate of tislelizumab combined with GX regimen and tislelizumab combined with GP regimen based on the ITT analysis set evaluated by the researchers according to RECISTv1.1. | up to approximately 3 years
  Complete remission rate+ partial remission rate

OTHER OUTCOMES:
To compare the duration of response of R/M NPC patients treated with tislelizumab combined with GX regimen and tislelizumab combined with GP regimen based on the intention-to-treat (ITT) analysis set evaluated by the researchers according to RECISTv1.1. | up to approximately 3 years
  Time from the date of first partial remission or complete remission to the date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
To compare the overall survival (OS) of R/M NPC patients treated with tislelizumab combined with GX regimen and tislelizumab combined with GP regimen based on the intention-to-treat (ITT) analysis set evaluated by the researchers according to RECISTv1.1. | up to approximately 3 years
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.
To compare the safety and tolerance of R/M NPC patients treated with tislelizumab combined with GX regimen and tislelizumab combined with GP regimen based on the intention-to-treat (ITT) analysis set evaluated by the researchers according to RECISTv1.1. | up to approximately 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided